CLINICAL TRIAL: NCT02398032
Title: CPAP Effect on Nocturnal Evolution of Chemosensitivity Determinants in Sleep Apnea-hypopnea Patients With Isolated Nocturnal Hypertension or Day-nigh Sustained Hypertension
Brief Title: CPAP in SAHS Patients With Hypertension
Acronym: SAHS2-3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Francisco Garcia-Rio, MD, Hospital Universitario La Paz
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 99/0252
Record Dates: First submitted 2013-04-01; First posted 2015-03-25 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Sleep Apnea Syndromes; Hypertension
Keywords: sleep apnea; hypertension; mechanosensitivity; chemosensitivity; adhesion factors
MeSH Terms: conditions — Sleep Apnea Syndromes; Hypertension | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP nasal (Experimental): Nasal continuous positive airway pressure, during the night
  Interventions: Device: CPAP nasal
- sham CPAP nasal (Sham Comparator): Nasal sham continuous positive airway pressure, during the night
  Interventions: Device: sham CPAP nasal

INTERVENTIONS:
Device: CPAP nasal — During the night
  Other Names: Nocturnal support with continuous positive airway pressure
  Arms: CPAP nasal
Device: sham CPAP nasal — During the night
  Other Names: sham CPAP
  Arms: sham CPAP nasal

SUMMARY:
Study objective: To assess the nocturnal changes in mechanosensitivity and chemosensitivity in hypertensive sleep apnea-hypopnea syndrome (SAHS) patients and in SAHS patients with isolated nocturnal hypertension. To value the continuous positive airway pressure (CPAP) effect on these parameters.

Design: Controlled cross-over longitudinal study. Settings: Madrid metropolitan area. Patients: Day-night sustained hypertensive and isolated nocturnal hypertensive patients with SAHS without previous treatment. At least 30 patients are needed.

Interventions: Patients will allocate in each treatment arm (CPAP vs. sham CPAP) during three months. Explorations will perform before and immediately after sleep at 0-, 3-, and 6-months of trial.

Measurements: 24-h urinary catecholamine, local vascular factors, angiotensin and aldosterone levels. Diaphragmatic tension-time index, metabolic rate, hypoxic withdrawal test, and ventilatory and inspiratory neural drive responses to progressive isocapnic hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Recent diagnosis of sleep apnea-hypopnea syndrome with an apnea-hypopnea index (AHI) > 10 h-1
* No previous treatment for SAHS or hypertension
* Diagnosis by 24-h ambulatory monitoring of blood pressure (AMBP) of isolated nocturnal hypertension (nighttime blood pressure of ≥120 mm Hg systolic or 70 mm Hg diastolic and a daytime blood pressure <135/85 mm Hg) or day-night sustained hypertension (nighttime blood pressure of ≥120 mm Hg or 70 mm Hg diastolic and a daytime blood pressure of ≥135 mm Hg systolic).

Exclusion Criteria:

* Severe hypertension (> 180/120 mmHg).
* Previous diagnosis of secondary hypertension.
* Myocardial infarction or stroke in the last three months.
* Severe diurnal sleepiness (Epworth score > 15)
* Previous diagnosis of chronic obstructive pulmonary disease, asthma, bronchiectasis, lung cancer, restrictive lung disease, chest wall disease or thoracic surgery.
* Previous diagnosis or clinical evidence of heart disease, neuromuscular disease or thyroid dysfunction.
* Morbid obesity (BMI > 40 Kg/m2)
* Respiratory infection in the last two months.
* Treatment with theophylline or systemic corticosteroids in the last two years.
* Excessive alcohol intake (>40 g/day)
* Absence of social or familiar support.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Effect of CPAP on the night-morning change in the withdrawal response and in the ventilatory and central drive responses to progressive isocapnic hypoxia. | 3 months
  To compare the effect of three months of CPAP therapy versus sham CPAP on the night-morning (pre- vs. post-sleep) change in the withdrawal response (decrease in ventilation caused by two breaths of 100% oxygen, %ΔV'I) and in the ventilatory and inspiratory neural drive responses to progressive isocapnic hypoxia (ΔV'I/arterial oxygen saturation (SaO2)/body surface area (BSA)] and Δ occlusion pressure at 0.1 s (P0.1)/arterial oxygen saturation (SaO2), respectively).

SECONDARY OUTCOMES:
CPAP effect on the night-morning change in the sniff diaphragmatic tension-time index | 3 months
  To compare the effect of three months of CPAP therapy versus sham CPAP on the night-morning (pre- vs. post-sleep) change in the sniff diaphragmatic tension-time index (TTdi)
CPAP effect on blood pressure | 3 months
  To compare the effect of three months of CPAP therapy on the blood pressure in SAHS patients with isolated nocturnal hypertension and SAHS patients with day-nigh sustained hypertension
CPAP effect on the serum levels of endothelin-1 and vascular endothelial cell adhesion molecule (VCAM)-1 | 3 months
  To compare the effect of three months of CPAP therapy versus sham CPAP on the serum levels of endothelin-1 and VCAM-1 in SAHS patients with isolated nocturnal hypertension and SAHS patients with day-nigh sustained hypertension
CPAP effect on the night-morning change in the rest metabolic rate | 3 months
  To compare the effect of three months of CPAP therapy versus sham CPAP on the night-morning (pre- vs. post-sleep) change in the rest metabolic rate (carbon dioxide production/oxygen uptake ratio, RER)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Garcia-Rio, MD, Principal Investigator — Hospital Universitario La Paz, IdiPAZ
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Casitas R, Martinez-Ceron E, Galera R, Cubillos-Zapata C, Gonzalez-Villalba MJ, Fernandez-Navarro I, Sanchez B, Garcia-Sanchez A, Zamarron E, Garcia-Rio F. The effect of treatment for sleep apnoea on determinants of blood pressure control. Eur Respir J. 2017 Nov 16;50(5):1701261. doi: 10.1183/13993003.01261-2017. Print 2017 Nov. PMID 29146604